CLINICAL TRIAL: NCT01296217
Title: "Evaluation of the Sentinel Lymph Node Technic of the Prostate by Laparoscopy"
Brief Title: Sentinel Lymph Node Detection in Prostate Surgery by Laparoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre René Gauducheau (Other)
Allocation: Not Applicable | Model: Single Group
Other Study IDs: BRD 07/11-M
Record Dates: First submitted 2011-02-11; First posted 2011-02-15 (Estimated); Last update posted 2011-03-04 (Estimated); Status verified 2011-02

CONDITIONS: Prostatic Neoplasms
Keywords: Patients with infiltrant prostatic carcinoma
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lymph nod detection (Experimental)
  Interventions: Procedure: lymph nod detection

INTERVENTIONS:
Procedure: lymph nod detection

SUMMARY:
In this study the investigators want to determine if the detection of lymph node is applicable in prostatectomy by laparoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years
* Diagnosis of invasive cancer of the prostate (T1 or T2 or T3)
* PSA ≥ 4,
* Gleason ≥ 6
* No treatment prior to surgery
* Indication of lymphadenectomy by coeliscopique
* ECOG or Karnofsky index 2
* Patient information and signed informed consent

Exclusion Criteria:

* neoadjuvant hormone therapy
* Interventions prior pelvic
* Patients who received anterior resection of part of prostate
* Patient or denied having an altered mental status
* Any contre indication to laparoscopy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)

PRIMARY OUTCOMES:
detection rate and false-negative rate for the sentinel lymph node detection | The day of at laparoscopy (Day 1)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre René Gauducheau, Nantes, France